CLINICAL TRIAL: NCT02964468
Title: Multicenter Dose-escalation Trial of Radiotherapy in Patients With Locally Advanced Rectal Cancer
Brief Title: Dose-escalation Trial of Preoperative Radiotherapy and Concurrent Chemotherapy in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Responsible Party: Principal Investigator, Fernando Campos, Doctor, Grupo de Investigación Clínica en Oncología Radioterapia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTRC--001
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Rectal Cancer; IMRT; Radiation Dose Escalation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment with IMRT Dose Escalation (Experimental): Dose Escalation Intensity Modulated Radiotherapy treatment
  Interventions: Radiation: Dose Escalation Intensity Modulated Radiotherapy treatment
- Treatment with 3DCRT (Active Comparator): 3DCRT treatment (sequential boost)
  Interventions: Radiation: 3DCRT treatment (sequential boost)

INTERVENTIONS:
Radiation: 3DCRT treatment (sequential boost) — Radiotherapy:
  3DCRT treatment (sequential boost) 25 fractions fraction 1,8Gy by administering a total dose of 45 Gy on tumor and lymph nodes and lymph node chains more pelvic margin determined according to protocol.
  3 fractions fraction 1,8Gy by sequentially administering an additional dose of tumor and lymph nodes 5,4Gy on more margin.
  Chemotherapy:
  According to routine clinical practice of the participating centers.
  Arms: Treatment with 3DCRT
Radiation: Dose Escalation Intensity Modulated Radiotherapy treatment — Radiotherapy:
  IMRT treatment (concomitant boost technique) 25 fractions fraction 2,15Gy by administering a total dose of tumor and lymph nodes 53,75Gy on more margin. Simultaneously we will proceed to the irradiation of pelvic lymph node chains according to protocol, a division of 1,8Gy per session until a total dose of 45 Gy.
  Chemotherapy:
  According to routine clinical practice of the participating centers.
  Arms: Treatment with IMRT Dose Escalation

SUMMARY:
The aim of this study is to evaluate the increase of radiation dose administered in patients diagnosed with locally advanced rectal cancer in terms of ypRC with tolerable toxicity, using IMRT (concomitant boost technique).

DETAILED DESCRIPTION:
The hypothesis that arises is an improvement in the proportion of pathological complete responses, resulting therapeutic gain, as a result of a higher dose of radiation delivered to the tumor volume without incurring a higher gastrointestinal toxicity to the patient or surgical complications later, thanks to the use of intensity modulated radiotherapy (concomitant boost technique) that allows us to significantly reduce the administered dose organs at risk.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of adenocarcinoma of the rectum
* Clinically determined to be stage T3 or T4,N0-N2, and M0 -staged by MRI or transrectal ultrasound of the rectum
* Patients who are medically operable and who have resectable adenocarcinoma of the rectum at least <11cm from the anal verge
* Adequate liver/renal and haematological function.
* Eastern Cooperative Oncology Group (ECOG) performance 0-2
* Age ≥ 18 years
* Full blood count obtained within 2 weeks prior to registration on study, with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Haemoglobin ≥ 8.0 g/dl
  * Serum creatinine within normal institutional limits
  * Bilirubin within normal institutional limits
  * AST and ALT < 2.5 x the IULN
* Patient must sign study specific informed consent prior to study entry

Exclusion Criteria:

* Prior systemic chemotherapy for colorectal cancer; note that prior chemotherapy for a different cancer is allowable.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Any evidence of distant metastases (M1)
* A synchronous primary colon carcinoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-05 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | Through study completion, an average of 2 years
  Pathologic evaluation of the surgical specimen as assessed by Mandard Tumor regression scoring
Gastrointestinal toxicity | Two years
  Gastrointestinal adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Tumor regression grade | Through study completion, an average of two years
  Pathologic evaluation of the surgical specimen
Disease free survival | Three years
Overall survival | Five years
Acute Toxicity | Two years
  Acute Toxicity including anorexia, nausea, vomiting, diarrhoea, dermatitis proctitis, urinary frequency/urgency as per common toxicity criteria V4.03
Quality of Life during the treatment | Three years after the study completion
  Assessed by EORTC QLQC30-CR29 questionnaries

CONTACTS AND LOCATIONS:
Overall Officials: Fernando López Campos, Investigator, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (9):
- Spain (9):
  - Hospital General de Elche, Elche, Alicante
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón
  - Hospital Universitario Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No